CLINICAL TRIAL: NCT02946385
Title: A Phase 2b Open-Label Multi-Center Study Assessing the Immunological Persistence of Antibodies at Approximately 2 Years After the Last Meningococcal Vaccination in Study V102_15 (NCT02212457) and the Response to a Booster Dose of GSK MenABCWY or Meningococcal Serogroup B Vaccines, in Healthy Adolescents
Brief Title: Study to Assess the Immunological Long-term Persistence of Antibodies (Abs) 2 Years After GlaxoSmithKline (GSK) Meningococcal ABCWY Vaccination in the V102_15 (NCT02212457) and Response to a Booster in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205613; V102_15E1 (Other: Novartis); 2016-002230-69 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Infections, Meningococcal
Keywords: meningococcal disease; meningitis; booster; antibody persistence
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ABCWY_ 0_2 Group (Experimental): Subjects who received 2 doses of MenABCWY vaccine at Month 0 and Month 2 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
  Interventions: Biological: Meningococcal ABCWY Vaccine
- ABCWY_0_2_6 Group (Experimental): Subjects who received 3 doses of MenABCWY vaccine at Month 0, Month 2 and Month 6 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
  Interventions: Biological: Meningococcal ABCWY Vaccine
- B_0_2 Group (Experimental): Subjects who received 2 doses of rMenB+OMV vaccine at Month 0 and Month 2 in study V102_15 (NCT02212457), and will receive 1 dose of rMenB+OMV in this extension study
  Interventions: Biological: Meningococcal B Recombinant vaccine
- ABCWY_ 0_6 Group (Experimental): Subjects who received 2 doses of MenABCWY vaccine at Month 0 and Month 6 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
  Interventions: Biological: Meningococcal ABCWY Vaccine
- ABCWY Naive Group (Active Comparator): Subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study (NCT02212457), and will receive 2 doses of MenABCWY in this extension study
  Interventions: Biological: Meningococcal ABCWY Vaccine
- rMenB+OMV Naive Group (Active Comparator): Subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study (NCT02212457), and will receive 2 doses of rMenB+OMV in this extension study
  Interventions: Biological: Meningococcal B Recombinant vaccine

INTERVENTIONS:
Biological: Meningococcal ABCWY Vaccine — Intramuscular injection of one booster dose at Day 1 to follow-on subjects in the ABCWY_ 0_2 Group, ABCWY_ 0_2_6 Group and ABCWY_ 0_6 Group, primed with 2 or 3 doses of the study vaccine and 2 doses at Days 1 and 61 to naïve subjects in the ABCWY naïve group.
  Other Names: MenABCWY
  Arms: ABCWY Naive Group; ABCWY_ 0_2 Group; ABCWY_ 0_6 Group; ABCWY_0_2_6 Group
Biological: Meningococcal B Recombinant vaccine — Intramuscular injection of one booster dose of the rMenB+OMV vaccine to subjects in the B_0_2 group, primed with 2 doses of the vaccine and intramuscular injection of 2 doses at Days 1 and 61 in the deltoid area of the non-dominant arm to naïve subjects in the rMenB+OMV Naïve group.
  Other Names: rMenB+OMV
  Arms: B_0_2 Group; rMenB+OMV Naive Group

SUMMARY:
The purpose of this study is to compare the persistence of 2 or 3 doses of the GSK MenABCWY vaccine, or 2 doses of GSK rMenB+OMV vaccine (Bexsero) administered to healthy adolescents at approximately 24 months after the last meningococcal vaccination in the parent study V102_15(NCT02212457), compared with baseline antibody levels in vaccine naïve subjects at similar age at enrolment.

DETAILED DESCRIPTION:
Naive subjects will be randomized 1:1 to receive MenABCWY or rMenB+OMV at Day 1. No randomization to treatment arm for follow-on subjects is required as vaccine groups remain the same as in the parent study V102_15 (NCT02212457).

Response to a booster dose of MenABCWY vaccine will also be assessed in follow-on subjects who received 2 or 3 doses of MenABCWY (at 0.2-, 0,.6- or 0,.2,.6-month schedules) in the parent study, and will be compared with responses to a single dose of MenABCWY in naive subjects (subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study).

Response to a booster dose of GSK Meningococcal B Recombinant vaccine (rMenB+OMV) will be assessed in subjects who received 2 doses of rMenB+OMV (at 0, 2-month schedule) in the parent study, and will be compared with responses to a single dose of rMenB+OMV in naive subjects.

ELIGIBILITY:
Inclusion Criteria:

Follow-on Participants

* Subjects from Finland and Poland previously enrolled in study V102_15 (NCT02212457) who have received all planned meningococcal vaccinations in the study
* Who have not received any additional meningococcal vaccination since the last meningococcal vaccination administered in the parent trial.
* Who have given written informed consent or assent after the nature of the study has been explained according to local regulatory requirements, prior to study entry. If the subject is under age 18 at the time of enrollment, the parent(s)/ legal guardian(s) of the subject should have given their written consent.
* Individuals of who the investigator believes can and will comply with the requirements of the protocol.
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Naive Group

* Male and female individuals of similar age (approximately 12-20 years) to follow-on subjects from V102_15 (NCT02212457) trial.
* Who have not received any meningococcal vaccination since birth
* Individuals who have given their written informed consent or assent after the nature of the study has been explained according to local regulatory requirements, prior to study entry. If the subject is under age 18 at the time of enrollment, the parent(s)/ legal guardian(s) of the subject should have given their written consent.
* Individuals of who the investigator believes can and will comply with the requirements of the protocol.
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

Follow-on Participants:

* Follow-on individuals not eligible to be enrolled in the study are those with:
* History of any meningococcal vaccine administration since last meningococcal vaccination administered in V102_15 (NCT02212457) parent study.
* Current or previous, confirmed or suspected disease caused by N. meningitidis, since termination from parent study.
* Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment.
* If the subject is female of childbearing potential, sexually active, and has not used any of the acceptable contraceptive methods for at least 2 months prior to study entry and for the duration of the trial.
* Pregnancy or breast-feeding
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component including diphtheria toxoid (CRM197) and latex.
* Progressive, unstable or uncontrolled clinical conditions.
* Any confirmed or suspected condition with impaired/altered function of immune system.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to the study vaccination or planned use throughout the study period. (For corticosteroids, this means prednisone, or equivalent, ≥ 20 mg/day. Inhaled, intranasal and topical steroids are allowed).
* Administration of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the 3 months prior to study enrolment.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Administration of any vaccine within 14 days or 28 days prior to enrollment in the study, or within 7 days after vaccination in the study.
* Clinical conditions representing a contraindication to intramuscular vaccination and/or blood draws.
* Who have received systemic antibiotic treatment within 3 days prior to any blood draw
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.

Naive Individuals

* Naive individuals not eligible to be enrolled in the study are those with:
* History of any meningococcal vaccine administration since birth.
* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrollment.
* If the subject is female of childbearing potential, sexually active, and has not used any of the acceptable contraceptive methods for at least 2 months prior to study entry and for the duration of the trial.
* Pregnancy or breast-feeding.
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any vaccine component including diphtheria toxoid (CRM197) and latex.
* Progressive, unstable or uncontrolled clinical conditions.
* Any confirmed or suspected condition with impaired/altered function of immune system.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 30 days prior to the study enrolment. (For corticosteroids, this means prednisone, or equivalent, ≥ 20 mg/kg/day. Inhaled, intranasal and topical steroids are allowed).
* Administration of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months or planned use throughout the study period.
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
* Individuals who are part of study personnel or close family members conducting this study.
* Administration of any vaccine within 14 days or 28 days prior to enrollment in the study, or within 7 days after first vaccination, and/or planned use of any vaccine 7 days prior to and 7 days after second vaccination.
* Clinical conditions representing a contraindication to intramuscular vaccination and/or blood draws.
* Who have received systemic antibiotic treatment within 3 days prior to any blood draw
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 604 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects enrolled in the study started the study.
Pre-assignment Details: Participant flow,baseline characteristics & immunogenicity analyses were performed on "randomized" population & Safety analysis on "treated" population.2 subjects from Naïve_ABCWY group received rMenB+OMV vaccine & not MenABCWY.Hence,number of subjects analyzed in Naïve_B & Naive_ABCWY groups in treated population differ from randomized population
Groups:
- B_0_2: Subjects who received 2 doses of rMenB+OMV vaccine at Month 0 and Month 2 in study V102_15 (NCT02212457), and will receive 1 dose of rMenB+OMV in this extension study
- ABCWY_0_2: Subjects who received 2 doses of MenABCWY vaccine at Month 0 and Month 2 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
- Naive_B: Subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study (NCT02212457), and will receive 2 doses of rMenB+OMV in this extension study
- ABCWY_0_6: Subjects who received 2 doses of MenABCWY vaccine at Month 0 and Month 6 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
- Naive_ABCWY: Subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study (NCT02212457), and will receive 2 doses of MenABCWY in this extension study
- ABCWY_0_2_6: Subjects who received 3 doses of MenABCWY vaccine at Month 0, Month 2 and Month 6 in study V102_15 (NCT02212457), and will receive 1 dose of MenABCWY in this extension study
Period: Overall Study
Arm/Group | B_0_2 | ABCWY_0_2 | Naive_B | ABCWY_0_6 | Naive_ABCWY | ABCWY_0_2_6
Started | 126 | 127 | 99 | 74 | 101 | 77
Completed | 126 | 127 | 96 | 74 | 99 | 76
Not Completed | 0 | 0 | 3 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | B_0_2 | ABCWY_0_2 | Naive_B | ABCWY_0_6 | Naive_ABCWY | ABCWY_0_2_6 | TOTAL
Number analyzed (Participants) | 126 | 127 | 99 | 74 | 101 | 77 | 604
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.8 (3.06) | 16.6 (3.15) | 16.2 (2.8) | 17.3 (2.96) | 16.5 (2.78) | 17.1 (2.98) | 16.7 (2.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 69 | 58 | 44 | 60 | 50 | 363
  Male | 44 | 58 | 41 | 30 | 41 | 27 | 241
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ASIAN | 0 | 0 | 0 | 0 | 0 | 1 | 1
  OTHER | 0 | 0 | 2 | 1 | 0 | 1 | 4
  WHITE | 126 | 127 | 97 | 73 | 100 | 75 | 598

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA Titers ≥LLOQ Against 4 Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y at 24 Months After Last Meningococcal Vaccination in Follow-on Subjects in V102_15 and at Day 1 in Naive Subjects
Description: The immunogenicity of MenABCWY or rMenB+OMV vaccines, is measured as the percentage of subjects with High-Throughput Human Serum Bactericidal Assay (HT-hSBA) titers greater or equal than (≥) Lower limit of quantification (LLOQ) against N. meningitidis serogroup B test strains and serogroups A,C, W and Y. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: At 24 months after the last meningococcal vaccination for all follow-on subjects and at Day 1 in the extension study for naive subjects
Population: Subjects in full analysis set(FAS) persistence(24 months after last vaccination in V102_15/Day 1)who were randomized(if naive) & provided evaluable serum sample with hSBA results for atleast 1 serogroup B test strain/serogroups A,C,W/Y at Day 1 in extension study.Subjects in group B_0_2 did not receive MenACWY vaccination in the parent study
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Naive_ALL: Subjects who are meningococcal vaccine-naive and of similar age to subjects enrolled from the parent study (NCT02212457), and will receive 2 doses of MenABCWY or rMenB+OMV in this extension study
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ALL
Number analyzed (Participants) | 127 | 75 | 74 | 125 | 198
Percentage of subjects
  Meningitis B M14459 Ab: number analyzed (Participants) | 121 | 74 | 72 | 123 | 198
  Meningitis B M14459 Ab | 18 [11.8 to 26.2] | 16 [8.7 to 26.6] | 25 [15.5 to 36.6] | 17 [10.9 to 24.9] | 5 [2.1 to 8.5]
  Meningitis B 96217 Ab: number analyzed (Participants) | 127 | 74 | 74 | 124 | 198
  Meningitis B 96217 Ab | 71 [62.1 to 78.6] | 81 [70.3 to 89.3] | 73 [61.4 to 82.6] | 81 [73.5 to 87.9] | 34 [27.3 to 40.9]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 127 | 75 | 74 | 124 | 198
  Meningitis B NZ98/254 Ab | 16 [9.9 to 23.3] | 15 [7.6 to 24.7] | 18 [9.7 to 28.2] | 15 [9.5 to 22.9] | 3 [0.8 to 5.8]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 126 | 75 | 73 | 125 | 196
  Meningitis B M07-0241084 Ab | 29 [21.6 to 38.1] | 31 [20.5 to 42.4] | 36 [24.7 to 47.7] | 28 [20.3 to 36.7] | 17 [12.3 to 23.4]
  Meningitis A human Ab: number analyzed (Participants) | 125 | 72 | 74 | 0 | 99
  Meningitis A human Ab | 15 [9.4 to 22.7] | 25 [15.5 to 36.6] | 27 [17.4 to 38.6] |  | 3 [0.6 to 8.6]
  Meningitis C human Ab: number analyzed (Participants) | 127 | 74 | 74 | 0 | 100
  Meningitis C human Ab | 83 [75.8 to 89.5] | 86 [76.5 to 93.3] | 85 [75.0 to 92.3] |  | 32 [23.0 to 42.1]
  Meningitis W human Ab: number analyzed (Participants) | 127 | 75 | 72 | 0 | 98
  Meningitis W human Ab | 52 [42.9 to 60.9] | 73 [61.9 to 82.9] | 64 [51.7 to 74.9] |  | 27 [18.1 to 36.4]
  Meningitis Y human Ab: number analyzed (Participants) | 126 | 73 | 73 | 0 | 99
  Meningitis Y human Ab | 52 [43.3 to 61.3] | 75 [63.9 to 84.7] | 62 [49.5 to 72.8] |  | 7 [2.9 to 14.0]

2. Primary Outcome: hSBA GMTs Against Each of Four Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y at 24 Months After Last Meningococcal Vaccination in Follow-on Subjects in V102_15 and at Day 1 in Naive Subjects
Description: The immunogenicity of MenABCWY or rMenB+OMV vaccines, is measured as the HT-hSBA geometric mean titers (GMTs) against N. meningitidis serogroup B test strains and serogroups A,C, W and Y. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ALL
Number analyzed (Participants) | 127 | 75 | 74 | 125 | 198
Titers
  Meningitis B M14459 Ab: number analyzed (Participants) | 121 | 74 | 72 | 123 | 198
  Meningitis B M14459 Ab | 2.05 [1.68 to 2.50] | 2 [1.55 to 2.57] | 2.55 [1.98 to 3.30] | 2.02 [1.66 to 2.45] | 1.21 [1.04 to 1.42]
  Meningitis B 96217 Ab: number analyzed (Participants) | 127 | 74 | 74 | 124 | 198
  Meningitis B 96217 Ab | 13 [10 to 17] | 19 [14 to 27] | 15 [11 to 22] | 20 [15 to 26] | 3.63 [2.94 to 4.48]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 127 | 75 | 74 | 124 | 198
  Meningitis B NZ98/254 Ab | 1.78 [1.48 to 2.16] | 1.72 [1.34 to 2.19] | 2.1 [1.64 to 2.69] | 1.72 [1.42 to 2.08] | 1.1 [0.95 to 1.28]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 126 | 75 | 73 | 125 | 196
  Meningitis B M07-0241084 Ab | 3.95 [3.09 to 5.05] | 4.22 [3.07 to 5.80] | 5.2 [3.77 to 7.18] | 4.21 [3.29 to 5.38] | 2.27 [1.87 to 2.77]
  Meningitis A human Ab: number analyzed (Participants) | 125 | 72 | 74 | 0 | 99
  Meningitis A human Ab | 2.25 [1.72 to 2.95] | 4.52 [3.18 to 6.44] | 4.89 [3.45 to 6.94] |  | 1.21 [0.89 to 1.63]
  Meningitis C human Ab: number analyzed (Participants) | 127 | 74 | 74 | 0 | 100
  Meningitis C human Ab | 18 [14 to 23] | 29 [21 to 41] | 20 [14 to 28] |  | 2.92 [2.19 to 3.89]
  Meningitis W human Ab: number analyzed (Participants) | 127 | 75 | 72 | 0 | 98
  Meningitis W human Ab | 39 [29 to 51] | 53 [36 to 76] | 44 [30 to 64] |  | 6.32 [4.59 to 8.70]
  Meningitis Y human Ab: number analyzed (Participants) | 126 | 73 | 73 | 0 | 99
  Meningitis Y human Ab | 9.19 [6.85 to 12] | 29 [20 to 43] | 16 [11 to 24] |  | 1.52 [1.09 to 2.12]

3. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers ≥ LLOQ Against 4 Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y at Day 31 After MenABCWY Vaccination in V102_15E1
Description: The immunogenicity of MenABCWY vaccine, was measured as the percentages of subjects with HT-hSBA titers greater than or equal to (≥) Lower limit of quantification (LLOQ) against N. meningitidis serogroup B test strains and serogroups A,C, W and Y. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: Day 31: One month after a booster dose of MenABCWY given at 24 months after last MenABCWY vaccination in groups: ABCWY_0_2, ABCWY_0_6 and ABCWY_0_2_6 and after first dose of MenABCWY in Naive_ABCWY Group
Population: All subjects in the FAS immunogenicity (Day 31, after booster dose[follow-on]/first dose[naive]) who were randomized (if naive), received at least one study vaccination and provided evaluable serum sample with results for at least one serogroup B test strain or serogroups A, C, W or Y at Day 31 in the extension study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 77 | 73 | 100
Percentage of subjects
  Meningitis B M14459 Ab: number analyzed (Participants) | 126 | 75 | 73 | 100
  Meningitis B M14459 Ab | 87 [79.3 to 91.9] | 85 [75.3 to 92.4] | 95 [86.6 to 98.5] | 29 [20.4 to 38.9]
  Meningitis B 96217 Ab | 100 [97.1 to 100] | 100 [95.3 to 100] | 100 [95.1 to 100] | 62 [51.7 to 71.5]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 127 | 76 | 72 | 100
  Meningitis B NZ98/254 Ab | 69 [60.5 to 77.2] | 68 [56.7 to 78.6] | 81 [69.5 to 88.9] | 27 [18.6 to 36.8]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 126 | 77 | 73 | 100
  Meningitis B M07-0241084 Ab | 87 [79.3 to 91.9] | 84 [74.4 to 91.7] | 81 [69.9 to 89.1] | 30 [21.2 to 40.0]
  Meningitis A human Ab: number analyzed (Participants) | 125 | 77 | 73 | 98
  Meningitis A human Ab | 98 [94.3 to 99.81] | 100 [95.3 to 100] | 99 [92.6 to 99.97] | 55 [44.7 to 65.2]
  Meningitis C human Ab: number analyzed (Participants) | 127 | 75 | 73 | 100
  Meningitis C human Ab | 100 [97.1 to 100] | 100 [95.2 to 100] | 100 [95.1 to 100] | 91 [83.6 to 95.8]
  Meningitis W human Ab: number analyzed (Participants) | 124 | 74 | 73 | 100
  Meningitis W human Ab | 100 [97.1 to 100] | 100 [95.1 to 100] | 100 [95.1 to 100] | 78 [68.6 to 85.7]
  Meningitis Y human Ab: number analyzed (Participants) | 127 | 76 | 73 | 98
  Meningitis Y human Ab | 100 [97.1 to 100] | 100 [95.3 to 100] | 99 [92.6 to 99.97] | 71 [61.4 to 80.1]

4. Secondary Outcome: Percentages of Subjects With 4-Fold Increase in HT-hSBA Titers Against 4 Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y at Day 31 After MenABCWY Vaccination in V102_15E1
Description: The immunogenicity of MenABCWY vaccine, was measured as the percentages of subjects with 4-Fold Increase in HT-hSBA Titers against N. meningitidis serogroup B test strains and serogroups A,C, W and Y. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab. The 4-fold titer rise is defined as: a) for subjects with pre-vaccination hSBA titers ˂ LLOQ, a post-vaccination hSBA ≥ 4 LLOQ; b) for subjects with a pre-vaccination hSBA titers ≥ LLOQ, an increase of at least 4 times of the pre-vaccination hSBA.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 75 | 73 | 99
Percentage of subjects
  Meningitis B M14459 Ab: number analyzed (Participants) | 120 | 73 | 72 | 99
  Meningitis B M14459 Ab | 54 [44.8 to 63.3] | 49 [37.4 to 61.3] | 65 [53.1 to 76.1] | 8 [3.6 to 15.3]
  Meningitis B 96217 Ab: number analyzed (Participants) | 127 | 74 | 73 | 99
  Meningitis B 96217 Ab | 91 [84.1 to 95.0] | 95 [86.7 to 98.5] | 97 [90.5 to 99.67] | 17 [10.3 to 26.1]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 127 | 75 | 72 | 99
  Meningitis B NZ98/254 Ab | 22 [15.2 to 30.3] | 17 [9.6 to 27.8] | 14 [6.9 to 24.1] | 16 [9.5 to 24.9]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 125 | 75 | 72 | 99
  Meningitis B M07-0241084 Ab | 38 [29.1 to 46.7] | 19 [10.6 to 29.3] | 17 [8.9 to 27.3] | 11 [5.7 to 19.0]
  Meningitis A human Ab: number analyzed (Participants) | 123 | 72 | 73 | 97
  Meningitis A human Ab | 82 [74.2 to 88.4] | 83 [72.7 to 91.1] | 88 [77.9 to 94.2] | 23 [14.8 to 32.3]
  Meningitis C human Ab: number analyzed (Participants) | 127 | 74 | 73 | 99
  Meningitis C human Ab | 94 [88.0 to 97.2] | 86 [76.5 to 93.3] | 93 [84.7 to 97.7] | 54 [43.2 to 63.6]
  Meningitis W human Ab: number analyzed (Participants) | 124 | 72 | 71 | 97
  Meningitis W human Ab | 93 [86.7 to 96.6] | 92 [82.7 to 96.9] | 85 [74.0 to 92.0] | 36 [26.6 to 46.5]
  Meningitis Y human Ab: number analyzed (Participants) | 126 | 73 | 72 | 96
  Meningitis Y human Ab | 94 [87.9 to 97.2] | 89 [79.5 to 95.1] | 90 [81.0 to 96.0] | 46 [35.6 to 56.3]

5. Secondary Outcome: hSBA GMTs Against Each of Four Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y at Day 31 After MenABCWY Vaccination in V102_15E1
Description: The immunogenicity of MenABCWY vaccine, was measured as the HT-hSBA Geometric Mean Titers (GMTs) against N. meningitidis serogroup B test strains and serogroups A,C, W and Y . The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 77 | 73 | 100
Titers
  Meningitis B M14459 Ab: number analyzed (Participants) | 126 | 75 | 73 | 100
  Meningitis B M14459 Ab | 32 [25 to 41] | 30 [22 to 42] | 61 [44 to 85] | 3.12 [2.34 to 4.14]
  Meningitis B 96217 Ab | 580 [467 to 722] | 529 [400 to 700] | 544 [408 to 725] | 11 [8.25 to 13]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 127 | 76 | 72 | 100
  Meningitis B NZ98/254 Ab | 16 [12 to 21] | 13 [9.04 to 18] | 16 [12 to 23] | 3.14 [2.32 to 4.24]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 126 | 77 | 73 | 100
  Meningitis B M07-0241084 Ab | 32 [26 to 41] | 25 [18 to 33] | 21 [16 to 29] | 4.48 [3.47 to 5.78]
  Meningitis A human Ab: number analyzed (Participants) | 125 | 77 | 73 | 98
  Meningitis A human Ab | 271 [211 to 348] | 267 [194 to 367] | 340 [245 to 472] | 17 [13 to 22]
  Meningitis C human Ab: number analyzed (Participants) | 127 | 75 | 73 | 100
  Meningitis C human Ab | 628 [498 to 791] | 602 [446 to 812] | 529 [391 to 718] | 48 [37 to 62]
  Meningitis W human Ab: number analyzed (Participants) | 124 | 74 | 73 | 100
  Meningitis W human Ab | 1309 [1062 to 1614] | 1078 [823 to 1413] | 979 [746 to 1286] | 129 [102 to 162]
  Meningitis Y human Ab: number analyzed (Participants) | 127 | 76 | 73 | 98
  Meningitis Y human Ab | 616 [479 to 791] | 606 [439 to 836] | 578 [415 to 803] | 33 [25 to 44]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLOQ Against 4 Serogroup B Test Strains, and N. Meningitidis Serogroups A, C, W and Y at 24 Months At Days 1, 6, 31 in V102_15 Follow-on Subjects and at Day 1, 66, 91 in Naive Subjects, in MenABCWY Groups
Description: The immunogenicity of MenABCWY vaccine, was measured as the percentages of subjects with HT-hSBA titers greater or equal than (≥) Lower limit of quantification (LLOQ) against N. meningitidis serogroup B test strains and serogroups A,C, W and Y. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: At Day 1, Day 6 and 31(after booster dose of MenABCWY given at 24 months after last MenABCWY vaccination) in ABCWY_0_2, ABCWY_0_6 and ABCWY_0_2_6 groups and at Day 1, Day 66 and 91(i.e. day 6 and 1 month after dose 2 of MenABCWY) in Naive_ABCWY Group
Population: All subjects in FAS immunogenicity(Days 6 and 31, after booster [follow-on]/D66 and 91 after dose 2[naive]) who were randomized(if naive), received at least 1 study vaccination and provided evaluable results for at least 1 serogroup B strain or serogroups A, C, W, Y at D1, and at least at D6 or D31(follow-on)/D 66 or D91(naive) in extension study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 75 | 72 | 96
Percentage of subjects
  Meningitis B M14459 Ab, Day 1: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, Day 1 | 18 [12.0 to 26.6] | 17 [8.9 to 27.3] | 26 [16.0 to 37.6] | 6 [2.4 to 13.4]
  Meningitis B M14459 Ab, Day 6 Post: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, Day 6 Post | 64 [54.6 to 72.5] | 82 [71.1 to 90.0] | 89 [78.7 to 94.9] | 64 [53.3 to 73.5]
  Meningitis B M14459 Ab, One month Post: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, One month Post | 86 [78.1 to 91.5] | 85 [74.3 to 92.1] | 94 [86.0 to 98.4] | 72 [62.2 to 81.1]
  Meningitis B 96217 Ab, Day 1: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, Day 1 | 71 [62.4 to 78.9] | 81 [70.3 to 89.3] | 74 [61.9 to 83.3] | 32 [23.1 to 42.6]
  Meningitis B 96217 Ab, Day 6 Post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, Day 6 Post | 98 [94.3 to 99.81] | 100 [95.1 to 100.0] | 97 [90.3 to 99.66] | 91 [82.9 to 95.6]
  Meningitis B 96217 Ab, One month Post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, One month Post | 100 [97.1 to 100.0] | 100 [95.1 to 100.0] | 100 [95.0 to 100.0] | 98 [92.7 to 99.75]
  Meningitis B NZ98/254 Ab, Day 1: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, Day 1 | 16 [9.9 to 23.3] | 14 [6.7 to 23.5] | 18 [10.1 to 29.3] | 2 [0.26 to 7.5]
  Meningitis B NZ98/254 Ab, Day 6 Post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, Day 6 Post | 44 [35.3 to 53.2] | 53 [40.7 to 64.4] | 66 [54.0 to 77.0] | 56 [45.8 to 66.6]
  Meningitis B NZ98/254 Ab, One month Post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, One month Post | 69 [60.5 to 77.2] | 70 [58.5 to 80.3] | 80 [69.1 to 88.8] | 73 [63.3 to 82.0]
  Meningitis B M07-0241084 Ab, Day 1: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, Day 1 | 30 [22.0 to 38.7] | 31 [20.5 to 42.4] | 37 [25.5 to 48.9] | 18 [10.8 to 27.1]
  Meningitis B M07-0241084 Ab, Day 6 Post: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, Day 6 Post | 65 [55.4 to 72.9] | 72 [60.4 to 81.8] | 76 [64.5 to 85.4] | 55 [44.2 to 65.0]
  Meningitis B M07-0241084, One month Post: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084, One month Post | 86 [79.0 to 91.8] | 85 [75.3 to 92.4] | 80 [69.1 to 88.8] | 62 [51.6 to 71.9]
  Meningitis A human Ab, Day 1: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, Day 1 | 16 [9.6 to 23.2] | 25 [15.8 to 37.1] | 28 [17.9 to 39.6] | 3 [0.7 to 9.1]
  Meningitis A human Ab, Day 6 Post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, Day 6 Post | 88 [80.5 to 93.0] | 96 [88.1 to 99.1] | 89 [79.3 to 95.1] | 82 [72.4 to 89.0]
  Meningitis A human Ab, One month Post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, One month Post | 98 [94.2 to 99.80] | 100 [94.9 to 100.0] | 99 [92.5 to 99.96] | 94 [86.5 to 97.6]
  Meningitis C human Ab, Day 1: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, Day 1 | 83 [75.8 to 89.5] | 86 [76.5 to 93.3] | 86 [75.9 to 93.1] | 32 [22.4 to 41.9]
  Meningitis C human Ab, Day 6 Post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, Day 6 Post | 99 [95.7 to 99.98] | 100 [95.1 to 100.0] | 99 [92.5 to 99.96] | 99 [94.3 to 99.97]
  Meningitis C human Ab, One month Post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, One month Post | 100 [97.1 to 100.0] | 100 [95.1 to 100.0] | 100 [95.0 to 100.0] | 100 [96.2 to 100.0]
  Meningitis W human Ab, Day 1: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, Day 1 | 52 [42.8 to 61.2] | 73 [61.4 to 83.1] | 64 [51.3 to 75.0] | 27 [18.2 to 37.1]
  Meningitis W human Ab, Day 6 Post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, Day 6 Post | 99 [95.5 to 99.98] | 99 [92.4 to 99.96] | 97 [89.9 to 99.65] | 98 [92.4 to 99.74]
  Meningitis W human Ab, One month Post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, One month Post | 100 [97.0 to 100.0] | 100 [94.9 to 100.0] | 100 [94.8 to 100.0] | 98 [92.4 to 99.74]
  Meningitis Y human Ab, Day 1: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, Day 1 | 52 [42.9 to 61.0] | 76 [64.9 to 85.6] | 62 [49.7 to 73.2] | 7 [3.0 to 14.7]
  Meningitis Y human Ab, Day 6 Post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, Day 6 Post | 97 [92.0 to 99.1] | 100 [95.0 to 100.0] | 97 [90.2 to 99.66] | 95 [88.0 to 98.3]
  Meningitis Y human Ab, One month Post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, One month Post | 100 [97.1 to 100.0] | 100 [95.0 to 100.0] | 99 [92.4 to 99.96] | 95 [88.0 to 98.3]

7. Secondary Outcome: Percentages of Subjects With 4-Fold Increase in HT-hSBA Titers Against 4 Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y At Days 6, 31 in Follow-on Subjects in V102_15 and at Day 66, 91 in Naive Subjects, in MenABCWY Groups
Description: as for outcome 4
Time Frame: At Day 6 and 31(after booster dose of MenABCWY given at 24 months after last MenABCWY vaccination) in ABCWY_0_2, ABCWY_0_6 and ABCWY_0_2_6 groups and at Day 66 and 91(i.e. day 6 and 1 month after dose 2 of MenABCWY) in Naive_ABCWY Group
Population: All subjects in FAS immunogenicity(Days 6 and 31, after booster[follow-on]/D66 and 91 after dose 2[naive]) who were randomized(if naive), received at least 1 study vaccination and provided evaluable results for at least 1 serogroup B strain or serogroups A, C, W, Y at D1, and at least at D6 or D31(follow-on)/D 66 or D91(naive) in extension study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 75 | 72 | 96
Percentage of subjects
  Meningitis B M14459 Ab, Day 6 Post vacc: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, Day 6 Post vacc | 26 [18.4 to 34.9] | 36 [25.1 to 48.3] | 50 [37.8 to 62.2] | 30 [20.8 to 40.1]
  Meningitis B M14459 Ab, One month Post vacc: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, One month Post vacc | 55 [45.2 to 63.8] | 49 [36.7 to 60.7] | 64 [51.9 to 75.4] | 24 [16.2 to 34.4]
  Meningitis B 96217 Ab, Day 6 Post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, Day 6 Post | 86 [79.1 to 91.9] | 92 [83.2 to 97.0] | 85 [74.3 to 92.1] | 65 [54.2 to 74.1]
  Meningitis B 96217 Ab, One month Post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, One month Post | 90 [83.8 to 94.9] | 95 [86.7 to 98.5] | 97 [90.3 to 99.66] | 73 [62.9 to 81.5]
  Meningitis B NZ98/254 Ab, Day 6 Post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, Day 6 Post | 4 [1.3 to 8.9] | 8 [3.0 to 16.8] | 14 [7.0 to 24.4] | 24 [16.2 to 34.4]
  Meningitis B NZ98/254 Ab, One month Post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, One month Post | 22 [15.2 to 30.3] | 18 [9.7 to 28.2] | 14 [7.0 to 24.4] | 21 [13.5 to 30.9]
  Meningitis B M07-0241084 Ab, Day 6 Post: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, Day 6 Post | 14 [8.2 to 21.0] | 11 [4.7 to 19.9] | 8 [3.2 to 17.5] | 8 [3.7 to 15.9]
  Meningitis B M07-0241084, One month Post: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084, One month Post | 37 [28.6 to 46.2] | 19 [10.6 to 29.3] | 15 [8.0 to 26.0] | 16 [9.1 to 24.7]
  Meningitis A human Ab, Day 6 Post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, Day 6 Post | 66 [56.4 to 73.9] | 76 [64.5 to 85.4] | 75 [63.4 to 84.5] | 53 [42.1 to 63.1]
  Meningitis A human Ab, One month Post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, One month Post | 82 [74.0 to 88.3] | 85 [74.0 to 92.0] | 88 [77.6 to 94.1] | 46 [35.8 to 56.9]
  Meningitis C human Ab, Day 6 Post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, Day 6 Post | 88 [81.3 to 93.2] | 86 [76.5 to 93.3] | 78 [66.4 to 86.7] | 83 [74.1 to 90.1]
  Meningitis C human Ab, One month Post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, One month Post | 94 [88.0 to 97.2] | 86 [76.5 to 93.3] | 93 [84.5 to 97.7] | 91 [82.8 to 95.6]
  Meningitis W human Ab, Day 6 Post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, Day 6 Post | 80 [71.9 to 86.9] | 85 [74.0 to 92.0] | 75 [63.5 to 84.9] | 62 [51.7 to 72.2]
  Meningitis W human Ab, One month Post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, One month Post | 93 [86.3 to 96.5] | 92 [82.5 to 96.8] | 84 [73.3 to 91.8] | 71 [60.6 to 79.9]
  Meningitis Y human Ab, Day 6 Post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, Day 6 Post | 81 [72.8 to 87.3] | 85 [74.3 to 92.1] | 79 [67.6 to 87.7] | 78 [67.9 to 85.6]
  Meningitis Y human Ab, One month Post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, One month Post | 94 [87.8 to 97.2] | 89 [79.3 to 95.1] | 90 [80.7 to 95.9] | 83 [73.8 to 89.9]

8. Secondary Outcome: hSBA GMTs Against Each of Four Serogroup B Test Strains, and Against N. Meningitidis Serogroups A, C, W and Y At Days 1, 6, 31 in Follow-on Subjects in V102_15 and at Day 1, 66, 91 in Naive Subjects, in MenABCWY Groups
Description: as for outcome 5
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | Naive_ABCWY
Number analyzed (Participants) | 127 | 75 | 72 | 96
Titers
  Meningitis B M14459 Ab, Day 1: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, Day 1 | 2.08 [1.70 to 2.54] | 2.04 [1.58 to 2.64] | 2.62 [2.02 to 3.41] | 1.28 [1.02 to 1.61]
  Meningitis B M14459 Ab, Day 6 post: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, Day 6 post | 13 [9.77 to 18] | 21 [14 to 31] | 40 [27 to 58] | 10 [7.48 to 14]
  Meningitis B M14459 Ab, One month post: number analyzed (Participants) | 119 | 72 | 70 | 94
  Meningitis B M14459 Ab, One month post | 30 [24 to 39] | 30 [22 to 42] | 61 [44 to 84] | 14 [10 to 18]
  Meningitis B 96217 Ab, Day 1: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, Day 1 | 13 [10 to 17] | 19 [14 to 27] | 16 [11 to 23] | 3.12 [2.31 to 4.22]
  Meningitis B 96217 Ab, Day 6 post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, Day 6 post | 376 [287 to 493] | 486 [343 to 690] | 401 [281 to 571] | 70 [51 to 95]
  Meningitis B 96217 Ab, One month post: number analyzed (Participants) | 125 | 74 | 72 | 96
  Meningitis B 96217 Ab, One month post | 587 [496 to 695] | 524 [421 to 652] | 550 [440 to 687] | 94 [77 to 114]
  Meningitis B NZ98/254 Ab, Day 1: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, Day 1 | 1.78 [1.47 to 2.16] | 1.66 [1.30 to 2.14] | 2.17 [1.68 to 2.80] | 1.07 [0.85 to 1.33]
  Meningitis B NZ98/254 Ab, Day 6 post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, Day 6 post | 6.02 [4.58 to 7.92] | 7.63 [5.33 to 11] | 12 [8.56 to 18] | 8.95 [6.52 to 12]
  Meningitis B NZ98/254 Ab, One month post: number analyzed (Participants) | 127 | 74 | 71 | 94
  Meningitis B NZ98/254 Ab, One month post | 17 [13 to 21] | 14 [10 to 19] | 17 [12 to 23] | 14 [10 to 18]
  Meningitis B M07-0241084 Ab, Day 1: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, Day 1 | 3.97 [3.10 to 5.09] | 4.22 [3.07 to 5.80] | 5.3 [3.81 to 7.35] | 2.18 [1.64 to 2.89]
  Meningitis B M07-0241084 Ab, Day 6 post: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, Day 6 post | 14 [11 to 18] | 17 [12 to 24] | 16 [12 to 23] | 8.68 [6.52 to 12]
  Meningitis B M07-0241084 Ab, One month: number analyzed (Participants) | 124 | 75 | 71 | 95
  Meningitis B M07-0241084 Ab, One month | 32 [26 to 40] | 26 [20 to 34] | 22 [16 to 28] | 11 [8.60 to 14]
  Meningitis A human Ab, Day 1: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, Day 1 | 2.31 [1.75 to 3.04] | 4.53 [3.16 to 6.48] | 5.13 [3.59 to 7.34] | 1.22 [0.89 to 1.68]
  Meningitis A human Ab, Day 6 post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, Day 6 post | 137 [98 to 191] | 221 [143 to 341] | 229 [149 to 352] | 59 [41 to 87]
  Meningitis A human Ab, One month post: number analyzed (Participants) | 122 | 71 | 72 | 93
  Meningitis A human Ab, One month post | 270 [222 to 327] | 275 [213 to 354] | 340 [264 to 437] | 85 [68 to 106]
  Meningitis C human Ab, Day 1: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, Day 1 | 18 [14 to 23] | 29 [21 to 41] | 21 [15 to 29] | 2.91 [2.17 to 3.92]
  Meningitis C human Ab, Day 6 post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, Day 6 post | 524 [414 to 662] | 694 [511 to 942] | 520 [381 to 710] | 153 [117 to 200]
  Meningitis C human Ab, One month post: number analyzed (Participants) | 127 | 74 | 72 | 95
  Meningitis C human Ab, One month post | 628 [523 to 753] | 612 [482 to 776] | 539 [423 to 686] | 177 [143 to 218]
  Meningitis W human Ab, Day 1: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, Day 1 | 38 [28 to 51] | 51 [35 to 75] | 44 [30 to 65] | 6.25 [4.48 to 8.72]
  Meningitis W human Ab, Day 6 post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, Day 6 post | 820 [665 to 1011] | 993 [756 to 1304] | 916 [694 to 1208] | 279 [220 to 353]
  Meningitis W human Ab, One month post: number analyzed (Participants) | 121 | 71 | 69 | 93
  Meningitis W human Ab, One month post | 1345 [1142 to 1584] | 1050 [849 to 1299] | 999 [805 to 1240] | 298 [247 to 359]
  Meningitis Y human Ab, Day 1: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, Day 1 | 9.11 [6.77 to 12] | 31 [21 to 45] | 17 [12 to 25] | 1.54 [1.10 to 2.16]
  Meningitis Y human Ab, Day 6 post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, Day 6 post | 351 [274 to 449] | 606 [439 to 837] | 425 [307 to 589] | 145 [109 to 192]
  Meningitis Y human Ab, One month post: number analyzed (Participants) | 125 | 72 | 71 | 94
  Meningitis Y human Ab, One month post | 623 [517 to 750] | 646 [506 to 824] | 586 [458 to 750] | 129 [104 to 159]

9. Secondary Outcome: Percentages of Subjects With HT-hSBA Titers ≥ LLOQ Against 4 Serogroup B Test Strains at Day 31 After rMenB+OMV Vaccination in V102_15E1
Description: The immunogenicity of rMenB+OMV vaccine, was measured as the percentages of subjects with HT-hSBA titers greater or equal than (≥) Lower limit of quantification (LLOQ) against N. meningitidis serogroup B test strains. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: Day 31: One month after a booster dose of rMenB+OMV given at 24 months after last rMenB+OMVl vaccination in B_0_2 Group and after first dose of rMenB+OMV in Naive_B Group
Population: All subjects in the FAS immunogenicity (Day 31, after booster dose[follow-on]/first dose[naive]) who were randomized (if naive), received at least one study vaccination and provided evaluable serum sample with results for at least one serogroup B test strain at Day 31 in the extension study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 124 | 98
Percentage of subjects
  Meningitis B M14459 Ab: number analyzed (Participants) | 123 | 96
  Meningitis B M14459 Ab | 94 [88.6 to 97.7] | 28 [19.4 to 38.2]
  Meningitis B 96217 Ab | 100 [97.1 to 100.0] | 74 [64.7 to 82.8]
  Meningitis B NZ98/254 Ab | 87 [79.9 to 92.4] | 27 [18.1 to 36.4]
  Meningitis B M07-0241084 Ab | 95 [89.8 to 98.2] | 33 [23.5 to 42.9]

10. Secondary Outcome: Percentages of Subjects With 4-Fold Increase in HT-hSBA Titers Against 4 Serogroup B Test Strains at Day 31 After rMenB+OMV Vaccination in V102_15E1
Description: The immunogenicity of rMenB+OMV vaccine, was measured as the percentages of subjects with 4-Fold Increase in HT-hSBA Titers against N. meningitidis serogroup B test strains. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab. The 4-fold titer rise is defined as: a) for subjects with pre-vaccination hSBA titers ˂ LLOQ, a post-vaccination hSBA ≥ 4 LLOQ; b) for subjects with a pre-vaccination hSBA titers ≥ LLOQ, an increase of at least 4 times of the pre-vaccination hSBA.
Time Frame: Day 31: One month after a booster dose of rMenB+OMV given at 24 months after last rMenB+OMV vaccination in B_0_2 Group and after first dose of rMenB+OMV in Naive_B Group
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 123 | 97
Percentage of subjects
  Meningitis B M14459 Ab: number analyzed (Participants) | 120 | 95
  Meningitis B M14459 Ab | 67 [57.5 to 75.0] | 15 [8.3 to 23.5]
  Meningitis B 96217 Ab: number analyzed (Participants) | 122 | 97
  Meningitis B 96217 Ab | 97 [91.8 to 99.1] | 19 [11.4 to 27.7]
  Meningitis B NZ98/254 Ab: number analyzed (Participants) | 122 | 97
  Meningitis B NZ98/254 Ab | 40 [31.4 to 49.4] | 16 [9.7 to 25.4]
  Meningitis B M07-0241084 Ab: number analyzed (Participants) | 123 | 95
  Meningitis B M07-0241084 Ab | 53 [43.6 to 61.9] | 8 [3.7 to 15.9]

11. Secondary Outcome: hSBA GMTs Against Each of Four Serogroup B Test Strains, at Day 31 After rMenB+OMV Vaccination in V102_15E1
Description: The immunogenicity of rMenB+OMV vaccine, was measured as the HT-hSBA geometric mean titers (GMTs) against N. meningitidis serogroup B test strains. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: as for outcome 10
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 124 | 98
Titers
  Meningitis B M14459 Ab: number analyzed (Participants) | 123 | 96
  Meningitis B M14459 Ab | 50 [39 to 65] | 3.48 [2.60 to 4.65]
  Meningitis B 96217 Ab | 820 [658 to 1023] | 18 [14 to 23]
  Meningitis B NZ98/254 Ab | 27 [21 to 35] | 3.14 [2.32 to 4.26]
  Meningitis B M07-0241084 Ab | 59 [47 to 74] | 4.82 [3.72 to 6.24]

12. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLOQ Against 4 Serogroup B Test Strains at 24 Months At Days 1, 6, 31 in Follow-on Subjects in V102_15 and at Day 1, 66, 91 in Naive Subjects, in rMenB+OMV Groups
Description: as for outcome 9
Time Frame: At Day 1, at Day 6 and 31(after a booster dose of rMenB+OMV given at 24 months after last rMenB+OMV vaccination) in B_0_2 Group, and at Day 1, at Day 66 and 91(i.e. day 6 and 1 month after second dose of rMenB+OMV) in Naive_B Group
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 122 | 94
Percentage of subjects
  Meningitis B 96217 Ab, Day 1: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, Day 1 | 82 [73.8 to 88.2] | 36 [26.5 to 46.7]
  Meningitis B 96217 Ab, Day 6 Post: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, Day 6 Post | 98 [92.9 to 99.5] | 88 [80.0 to 94.0]
  Meningitis B 96217 Ab, One month Post: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, One month Post | 100 [97.0 to 100.0] | 98 [92.5 to 99.74]
  Meningitis B M07-0241084 Ab, Day 1: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084 Ab, Day 1 | 28 [20.1 to 36.7] | 16 [9.4 to 25.5]
  Meningitis B M07-0241084 Ab, Day 6 Post: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084 Ab, Day 6 Post | 70 [60.7 to 77.7] | 57 [45.8 to 66.8]
  Meningitis B M07-0241084, One month Post: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084, One month Post | 95 [89.6 to 98.2] | 72 [61.4 to 80.6]
  Meningitis B M14459 Ab, Day 1: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, Day 1 | 18 [11.3 to 25.7] | 3 [0.7 to 9.0]
  Meningitis B M14459 Ab, Day 6 Post: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, Day 6 Post | 70 [60.7 to 77.8] | 68 [57.7 to 77.3]
  Meningitis B M14459 Ab, One month Post: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, One month Post | 94 [88.3 to 97.6] | 78 [67.9 to 85.6]
  Meningitis B NZ98/254 Ab, Day 1: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, Day 1 | 16 [9.7 to 23.4] | 3 [0.7 to 9.0]
  Meningitis B NZ98/254 Ab, Day 6 Post: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, Day 6 Post | 49 [39.6 to 58.0] | 62 [51.1 to 71.5]
  Meningitis B NZ98/254 Ab, One month Post: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, One month Post | 87 [79.4 to 92.2] | 82 [72.6 to 89.1]

13. Secondary Outcome: Percentages of Subjects With 4-Fold Increase in HT-hSBA Titers Against 4 Serogroup B Test Strains At Days 6, 31 in Follow-on Subjects in V102_15 and at Day 66, 91 in Naive Subjects, in rMenB+OMV Groups
Description: as for outcome 10
Time Frame: At Day 6 and 31(after a booster dose of rMenB+OMV given at 24 months after last rMenB+OMV vaccination) in B_0_2 Group, and at Day 66 and 91(i.e. day 6 and 1 month after second dose of rMenB+OMV) in Naive_B Group
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 116 | 78
Percentage of subjects
  Meningitis B M14459 Ab, Day 6 Post: number analyzed (Participants) | 113 | 77
  Meningitis B M14459 Ab, Day 6 Post | 34 [25.0 to 43.1] | 22 [13.4 to 33.0]
  Meningitis B M14459 Ab, One month Post: number analyzed (Participants) | 113 | 77
  Meningitis B M14459 Ab, One month Post | 66 [56.9 to 75.0] | 31 [21.1 to 42.7]
  Meningitis B 96217 Ab, Day 6 Post: number analyzed (Participants) | 116 | 77
  Meningitis B 96217 Ab, Day 6 Post | 78 [69.9 to 85.5] | 69 [57.3 to 78.9]
  Meningitis B 96217 Ab, One month Post: number analyzed (Participants) | 116 | 77
  Meningitis B 96217 Ab, One month Post | 97 [92.6 to 99.5] | 81 [69.9 to 88.7]
  Meningitis B NZ98/254 Ab, Day 6 Post: number analyzed (Participants) | 115 | 78
  Meningitis B NZ98/254 Ab, Day 6 Post | 13 [7.5 to 20.6] | 21 [12.2 to 31.2]
  Meningitis B NZ98/254 Ab, One month Post: number analyzed (Participants) | 115 | 78
  Meningitis B NZ98/254 Ab, One month Post | 41 [31.8 to 50.4] | 41 [30.0 to 52.7]
  Meningitis B M07-0241084 Ab, Day 6 Post: number analyzed (Participants) | 116 | 76
  Meningitis B M07-0241084 Ab, Day 6 Post | 21 [13.7 to 29.2] | 14 [7.5 to 24.4]
  Meningitis B M07-0241084, One month Post: number analyzed (Participants) | 116 | 76
  Meningitis B M07-0241084, One month Post | 53 [43.1 to 61.9] | 24 [14.7 to 34.8]

14. Secondary Outcome: hSBA GMTs Against Each of Four Serogroup B Test Strains At Days 1, 6, 31 in Follow-on Subjects in V102_15 and at Day 1, 66, 91 in Naive Subjects, in rMenB+OMV Groups
Description: as for outcome 11
Time Frame: as for outcome 12
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | B_0_2 | Naive_B
Number analyzed (Participants) | 122 | 94
Titers
  Meningitis B M14459 Ab, Day 1: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, Day 1 | 2.04 [1.67 to 2.49] | 1.18 [0.94 to 1.47]
  Meningitis B M14459 Ab, Day 6 post: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, Day 6 post | 14 [11 to 19] | 12 [8.41 to 16]
  Meningitis B M14459 Ab, One month post: number analyzed (Participants) | 119 | 94
  Meningitis B M14459 Ab, One month post | 49 [38 to 63] | 16 [12 to 21]
  Meningitis B 96217 Ab, Day 1: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, Day 1 | 20 [15 to 26] | 4.38 [3.23 to 5.93]
  Meningitis B 96217 Ab, Day 6 post: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, Day 6 post | 341 [259 to 448] | 85 [63 to 116]
  Meningitis B 96217 Ab, One month post: number analyzed (Participants) | 121 | 94
  Meningitis B 96217 Ab, One month post | 822 [692 to 975] | 122 [100 to 148]
  Meningitis B NZ98/254 Ab, Day 1: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, Day 1 | 1.72 [1.41 to 2.09] | 1.15 [0.92 to 1.44]
  Meningitis B NZ98/254 Ab, Day 6 post: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, Day 6 post | 6.39 [4.83 to 8.45] | 9.38 [6.83 to 13]
  Meningitis B NZ98/254 Ab, One month post: number analyzed (Participants) | 121 | 94
  Meningitis B NZ98/254 Ab, One month post | 27 [21 to 34] | 22 [17 to 29]
  Meningitis B M07-0241084 Ab, Day 1: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084 Ab, Day 1 | 4.24 [3.30 to 5.45] | 2.36 [1.77 to 3.15]
  Meningitis B M07-0241084 Ab, Day 6 post: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084 Ab, Day 6 post | 17 [13 to 21] | 11 [8.54 to 15]
  Meningitis B M07-0241084 Ab, One month post: number analyzed (Participants) | 122 | 92
  Meningitis B M07-0241084 Ab, One month post | 59 [47 to 72] | 17 [13 to 22]

15. Secondary Outcome: Number of Subjects With Any Solicited Local or Systemic AEs and Other Indicators of Reactogenicity Within 30 Minutes After Vaccination
Description: Assessed solicited symptoms were Pain, erythema and induration. Assessed solicited systemic symptoms were Fatigue, headache, myalgia, arthralgia, loss of appetite, nausea, chills, and fever (body temperature ≥38.0°C).
Time Frame: within 30 minutes after vaccination at Day 1 (for all subjects) and also Day 61 (for naive subjects only)
Population: Analysis was done on subjects in Solicited Safety Set: all screened subjects who provided informed consent, demographic and/or other baseline screening measurements, regardless of the subject's randomization and vaccination status in the trial, received subject ID and study vaccination, and provided post-vaccination solicited adverse events data
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ABCWY | Naive_B
Number analyzed (Participants) | 127 | 77 | 74 | 126 | 99 | 101
Participants
  Local: Erythema: number analyzed (Participants) | 125 | 77 | 74 | 125 | 99 | 101
  Local: Erythema | 1 | 1 | 1 | 0 | 0 | 0
  Local: Induration: number analyzed (Participants) | 126 | 77 | 74 | 126 | 99 | 101
  Local: Induration | 0 | 1 | 0 | 0 | 0 | 0
  Local: Pain | 6 | 4 | 3 | 11 | 10 | 13
  Systemic: Arthralgia | 0 | 0 | 0 | 0 | 1 | 0
  Systemic: Chills | 0 | 0 | 0 | 0 | 0 | 0
  Systemic: Fatigue | 0 | 1 | 0 | 2 | 3 | 2
  Systemic: Fever | 0 | 0 | 0 | 0 | 0 | 0
  Systemic: Headache | 1 | 0 | 1 | 0 | 2 | 1
  Systemic: Loss Of Appetite | 0 | 0 | 0 | 0 | 1 | 0
  Systemic: Myalgia | 1 | 0 | 0 | 0 | 2 | 0
  Systemic: Nausea: number analyzed (Participants) | 127 | 77 | 74 | 125 | 99 | 101
  Systemic: Nausea | 1 | 0 | 0 | 1 | 0 | 2
  Indicator: Prevention Of Pain / Fever | 0 | 0 | 0 | 0 | 0 | 0
  Indicator: Treatment Of Pain / Fever | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Any Unsolicited AEs Within 30 Minutes After Vaccination
Description: An unsolicited adverse event is an adverse event that was not solicited and that was spontaneously communicated by a subject and/or parent/legal guardian who has signed the informed consent. Number of subjects reporting any unsolicited AE within 30 minutes after each vaccination. Note: unsolicited AEs within 30 minutes were not collected
Time Frame: Within 30 minutes after vaccination at Day 1 (for all subjects) and also Day 61 (for naive subjects only)
Population: Analysis was to be done on subjects in Unsolicited Safety Set but was not performed as AEs within 30 minutes after vaccination were not collected.
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ABCWY | Naive_B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects With Any Solicited Local or Systemic Adverse Events (AEs) and Other Indicators of Reactogenicity From Day 1 to Day 7.
Description: as for outcome 15
Time Frame: At Day 1 (6 hours) to Day 7 after vaccination at Day 1 (for all subjects) and Day 61 to Day 67 (for naive subjects only)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ABCWY | Naive_B
Number analyzed (Participants) | 127 | 77 | 74 | 126 | 99 | 101
Participants
  Local: Erythema | 22 | 10 | 14 | 22 | 23 | 20
  Local: Induration | 18 | 14 | 6 | 20 | 22 | 15
  Local: Pain | 108 | 67 | 64 | 115 | 95 | 93
  Systemic: Arthralgia | 12 | 5 | 9 | 15 | 19 | 17
  Systemic: Chills | 23 | 8 | 12 | 27 | 25 | 26
  Systemic: Fatigue | 58 | 33 | 31 | 64 | 59 | 55
  Systemic: Fever | 8 | 3 | 1 | 6 | 3 | 6
  Systemic: Headache | 55 | 19 | 28 | 61 | 61 | 45
  Systemic: Loss Of Appetite | 15 | 9 | 7 | 20 | 20 | 16
  Systemic: Myalgia | 26 | 13 | 14 | 22 | 26 | 21
  Systemic: Nausea | 13 | 8 | 8 | 24 | 20 | 19
  Indicator: Prevention Of Pain / Fever | 21 | 8 | 8 | 29 | 24 | 26
  Indicator: Treatment Of Pain / Fever | 37 | 18 | 19 | 56 | 47 | 39

18. Secondary Outcome: Number of Subjects With Unsolicited AEs, 30 Days After Any Vaccination
Description: An unsolicited adverse event is an adverse event that was not solicited and that was spontaneously communicated by a subject and/or parent/legal guardian who has signed the informed consent. Number of subjects reporting any unsolicited AE within 30 minutes after each vaccination.
Time Frame: From Day 1 to Day 31 for all subjects and Day 61 to Day 91 for naive subjects
Population: Analysis was done on subjects in Unsolicited Safety Set: all screened subjects who provided informed consent, demographic and/or other baseline screening measurements, regardless of subject's randomization and vaccination status in the trial, received subject ID and study vaccination, and provided post-vaccination unsolicited adverse events data
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ABCWY | Naive_B
Number analyzed (Participants) | 127 | 77 | 74 | 126 | 99 | 101
Participants | 27 | 12 | 10 | 26 | 40 | 36

19. Secondary Outcome: Number of Subjects With Any Serious AE (SAE), Medically Attended AEs (MAAEs), AEs Leading to Premature Withdrawal
Description: Serious adverse events (SAEs), medically attended adverse events and AEs leading to withdrawal are reported. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in one or more of the following: -Death, -Is life-threatening,-Required or prolonged hospitalization, -Persistent or significant disability/incapacity, -Congenital anomaly/or birth defect, -An important and significant medical event that may not be immediately life threatening or resulting in death or hospitalization but, based upon appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above.
Time Frame: During the entire study period (up to Day 181 for follow-on subjects and up to Day 241 for naive subjects)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | ABCWY_0_2 | ABCWY_0_2_6 | ABCWY_0_6 | B_0_2 | Naive_ABCWY | Naive_B
Number analyzed (Participants) | 127 | 77 | 74 | 126 | 99 | 101
Participants
  Any medically attended AE | 18 | 7 | 8 | 20 | 24 | 21
  Any serious AE | 0 | 0 | 0 | 2 | 0 | 1
  AEs leading to premature withdrawal | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7, and Unsolicited AEs from Day 1 to Day 30, after any vaccination. SAEs were collected throughout the entire study period (up to Day 181 for follow-on subjects and up to Day 241 for naive subjects).
Description: Safety analysis was performed on the treated population.
Arm/Group | B_0_2 | ABCWY_0_2 | Naive_B | ABCWY_0_6 | Naive_ABCWY | ABCWY_0_2_6
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/127 | 0/101 | 0/74 | 0/99 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/126 | 0/127 | 1/101 | 0/74 | 0/99 | 0/77
Other Adverse Events (participants affected / at risk) | 120/126 | 116/127 | 99/101 | 67/74 | 96/99 | 70/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B_0_2 (N=126) | ABCWY_0_2 (N=127) | Naive_B (N=101) | ABCWY_0_6 (N=74) | Naive_ABCWY (N=99) | ABCWY_0_2_6 (N=77)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B_0_2 (N=126) | ABCWY_0_2 (N=127) | Naive_B (N=101) | ABCWY_0_6 (N=74) | Naive_ABCWY (N=99) | ABCWY_0_2_6 (N=77)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (33) | 13 (21) | 17 (33) | 9 (18) | 20 (38) | 6 (9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 27 (50) | 23 (39) | 26 (62) | 12 (20) | 25 (51) | 8 (12)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (39) | 15 (15) | 16 (38) | 7 (13) | 20 (49) | 9 (11)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 3 (5) | 3 (3) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyssomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 64 (164) | 58 (114) | 55 (206) | 31 (77) | 59 (201) | 33 (67)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 62 (132) | 55 (96) | 46 (160) | 28 (64) | 62 (183) | 20 (41)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 59 (129) | 50 (100) | 49 (137) | 27 (67) | 45 (148) | 23 (53)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 40 (117) | 43 (107) | 43 (172) | 18 (51) | 46 (200) | 23 (58)
Injection site pain (General disorders) | 116 (421) | 108 (321) | 93 (683) | 64 (226) | 95 (593) | 67 (227)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine-triggered seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (42) | 26 (36) | 21 (40) | 14 (34) | 26 (57) | 13 (17)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 3 (4) | 1 (1) | 6 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 26 (39) | 13 (20) | 21 (39) | 8 (10) | 20 (39) | 8 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 8 (8) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 10 (11) | 6 (6) | 1 (1) | 5 (6) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal varicose veins (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal flattening (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8) | 11 (13) | 4 (4) | 6 (8) | 1 (1)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT02946385/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT02946385/SAP_001.pdf